CLINICAL TRIAL: NCT03085771
Title: Desferal Administration to Improve the Impaired Reaction to Hypoxia in Diabetes
Acronym: DESIRED
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Sergiu Catrina, Senior consultant / associated professor, Karolinska University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016/1925-31
Record Dates: First submitted 2017-03-07; First posted 2017-03-21 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Deferoxamine; Sodium Chloride; Isotonic Solutions

STUDY DESIGN:
Intervention Model Description: This is a randomised, double-blind, placebo-controlled, cross-over, single center study of patients with diabetes mellitus type 1 without chronic complications.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desferal treatment (Active Comparator): Patients will be randomized (by block randomization) to Desferal (DFO) treatment.
  Interventions: Drug: desferal
- Isotonic saline treatment (Placebo Comparator): Patients will be randomized (by block randomization) to isotonic saline treatment.
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: desferal — It is a blinded randomized cross-over study that investigates the efficacy of DFO (50mg/kg) given i.v before intermittent hypoxia (IH) to improve the cardiorespiratory and angiogenetic response in patients with diabetes.
  Other Names: deferoxamine
  Arms: Desferal treatment
Drug: Isotonic saline — It is a blinded randomized cross-over study that investigates the efficacy of isotonic saline given i.v before intermittent hypoxia (IH) to improve the cardiorespiratory and angiogenetic response in patients with diabetes.
  Other Names: Isotonic solution
  Arms: Isotonic saline treatment

SUMMARY:
The general aim of this study is to investigate the influence of systemic administration of Desferal (Deferoxamine [DFO]) on the response to hypoxic challenge in patients with diabetes mellitus (DM).

The investigation will elucidate if DFO can restore:

* the impaired angiogenetic response to hypoxia in patients with type 1 DM.
* the disturbed respiratory and cardiovascular regulation in response to hypoxia in patients with DM type 1

DETAILED DESCRIPTION:
Background Complications of diabetes represent the main concern for modern diabetes therapy, and it has become a priority to further characterize the pathophysiological mechanisms of these complications to ensure the development of novel rational therapeutic strategies.

Although the prolonged exposure of tissues to hyperglycemia is the primary causative factor for chronic diabetes complications, it has recently become increasingly evident that hypoxia also plays an important role in all diabetes complication. A low tissue concentration of oxygen in diabetes is the consequence of several mechanisms (e.g., deficient blood supply secondarily to micro- and macro-vascular disease, poor local oxygen diffusion secondarily to local edema or as a result of increased oxygen consumption).

Adaptive responses of the cells to hypoxia are mediated by Hypoxia-Inducible Factor 1 (HIF), which is a heterodimeric transcription factor, composed of two subunits (alfa and beta subunit) both constitutively expressed in mammalian cells. In normoxia, HIF-1α is continually degraded by the ubiquitin-proteasome system as a consequence of the oxygen-dependent hydroxylation of two key proline residues catalyzed by a group of enzymes called prolyl-hydroxylases (PHDs). Under hypoxia when the degradation pathway is suppressed and HIF-1α is stabilized, it translocates in the nucleus where it induces more than 800 genes that are

involved in angiogenesis, glycolytic energy metabolism, cell proliferation and survival that enable the cells to adapt to reduced oxygen availability. HIF-1 is central for expression of several angiogenic growth factors (ex. as Vascular Endothelial Growth Factor (VEGF), erythropoietin (EPO), and stromal cell-derived factor-1α (SDF-1α) and for endothelial progenitor cells (EPC) recruitment. Recently, it has been proposed that microRNAs (ex. mir210) also mediate a part of the HIF-1 functions.

PHDs that control the HIF 1 α stability and function are Fe 2+ and/or O2 -dependent enzymes and their activity could be inhibited by depleting the iron. Deferoxamine (DFO), which is an iron chelator induces therefore HIF-1α accumulation and hypoxia-response genes in normoxia both in vitro and in vivo being able to restore the repressed adaptative reaction to hypoxia different animal models of diabetes. DFO has been in clinical use for decades for treating excessive iron deposition secondary to different pathologies (thalassemia, myelosclerosis etc) and was used as pharmacological tool to induce HIF dependent responses.

In the last decade several pieces of evidence have gathered, point out that in diabetes there is a defective cellular response to hypoxia. An impaired hypoxia response is present in all tissues that develop complications both in animal models for diabetes and in patients with diabetes as a consequence of a defective HIF signaling. It is a direct effect of hyperglycemia that directly represses HIF stability and function at multiple levels.

The recently described impaired reaction to hypoxia in diabetes have potentially important consequences in acute hypoxic challenges as acute heart infarction, stroke, limb ischemia (known to have a worse prognosis in diabetes) but also in subtle regulation of cardiovascular and respiratory system as a consequence of autonomic neuropathy with potential severe prognostic effect on late cardiovascular events. Different studies have addressed the cardiovascular responses to intermittent hypoxia (IH) compared with normoxia exposure in patients with diabetes. In order to establish the appropriateness of the cardiovascular reaction to hypoxia in diabetes the cardiorespiratory and angiogenetic responses towards IH in patients with diabetes compared with matched non- diabetic control subjects has recently been investigated(HYKRAND ethical approval number 2015/1182-31/4). The preliminary results (not published) showed several defects in both acute and delayed reaction of the patients with diabetes compared with controls. The baroreflex sensitivity (BRS) which is a marker of cardiovascular risk and survival prognosis after cardiovascular events was decreased in patients with diabetes after IH compared with non-diabetic subjects. Both the Endothelial Precursors Cells (EPC) number and the levels of their main stimulator Stromal derived factor (SDF-1α) were decreased in in response to IH in diabetics compared with non- diabetic subjects confirming the worse capacity to repair ischemic lesions in diabetes.

The project proposed here investigate the potential of DFO (known to improve the HIF dependent hypoxic signaling) to reverse the impaired cardiorespiratory and angiogenetic response in diabetic patients.

Research design. It is a blinded randomized cross-over study that investigates the efficacy of DFO (50mg/kg) vs isotonic saline given i.v before intermittent hypoxia (IH) to improve the cardiorespiratory and angiogenetic response in patients with diabetes. IH will consist in five hypoxic periods (13% O2 inspired fraction of oxygen) each lasting 6 min, with five normoxic intervals of same duration (as used in HYKRAND study) in 30 patients with type 1 diabetes without clinical signs of any complication. The study will be performed during 4 days with minimum 2 months separation between the 2 admissions to ensure sufficient wash-out and to restore iron deposits.

Methods Study design This is a randomized, double blind study conducted in patients with diabetes type 1 without chronic complications.

Patients will be randomized (by block randomization) (httpps://www.sealedenvelope.com/ simple-randomiser/v1/lists) to (A) Desferal (DFO) treatment or (B) isotonic saline treatment.

Both the patients and the personnel will be blinded to the patient's treatment group.

Subjects will be advised to abstain from caffeinated beverages for 12 h and from alcohol for 36h prior to testing

Day 1: Baseline blood samples will be collected in the morning and afterwards the patients will receive Desferal (50 mg/kg) / Saline infusion s.c during 6hs. During the last hour of infusion the subjects will be exposed to intermittent hypoxia (IH). Blood samples and cardiovascular and respiratory (CR) measurements will be performed (as detailed below) immediately before and at several time points after IH.

Day 2: Blood samples will be collected in the morning. IH exposure consists of five hypoxic periods (13% O2 inspired fraction of oxygen) each lasting 6 min, with five normoxic intervals of same duration (totally 1 hour).

Day 1: blood pressure, heart rate and arterial oxygen saturation are continuously measured. In case of a decrease in oxygen saturation 80% or the occurrence of symptoms, hypoxia is discontinued until oxygen levels reached at least 80%. A technician regulates and control the breathing periods under supervision of a medical doctor in a way that the intervention could not be observed by the patient. Thereafter, three measurement sessions will be performed: immediately after (t2), after 3 h (t3), and after 6 h (t4). After t2, each patient obtained an individual meal according to diet requirement.

Cardiovascular and respiratory testing.

Assessment of baroreflex sensitivity. All patients will be tested in the supine position in a silent room at comfortable temperature. Before participants will be connected to a rebreathing circuit through a mouthpiece with an antibacterial filter, spontaneous breathing of room air at rest will be performed for 4 min in order to obtain baseline data.

During each condition, continuous measurement of oxygen saturation (SaO2) by a pulse oximeter and end-tidal CO2 (CO2-et) using a capnograph connected to a mouthpiece will be performed. Recordings of electrocardiogram will be performed by chest leads, and continuous noninvasive blood pressure will be recorded using the cuff method. Two belts (positioned around the chest and the abdomen) will monitor respiratory movements of the chest. A pneumotachograph will be connected to a differential pressure transducer and inserted in series to the expiratory component of the rebreathing system to measure airway flow.

The baroreflex sensitivity (BRS) will be measured during spontaneous breathing at each measurement session. Since previous studies did not document a better performance of one method over the others, the average of seven different methods: positive and negative sequences, the a-coefficient in the low- and high-frequency bands and its average, the transfer function technique, and the ratio of SDs of R-R interval and systolic blood pressure variabilities will be calculated. Besides BRS, SD of the R-R interval (SDNN) was applied to determine a global index of heart rate variability. This selection is done based on the fact that normal distribution is more pronounced in this variable compared with other indices of variability (e.g., variance).

Hypoxic ventilatory response (HVR) and hypercapnic ventilatory response (HCVR) will be evaluated to determine respiratory system activity.

Cardiovascular autonomic function will be determined performing four tests according to recent guidelines: deep-breathing, 30:15 ratio, Valsalva maneuver and systolic blood pressure response to standing. Cardiovascular autonomic neuropathy will be defined as the "presence of two or more abnormal tests".

The baroreflex sensitivity (BRS) will be evaluated before (t1), immediately after (t2), 3 h (t3), and 6 h (t4) after IH.

The angiogenetic potential will be evaluated at the same endpoints and after 24 H (Day N3) by measuring in serum relevant cytokines that are gene targets for HIF-1 (i.e. Vascular endothelial growth factor (AVEGFA), stromal cell-derived factor 1a (SDF-1a), erythropoietin etc.). The direct response of HIF signaling will be evaluated by the serum levels of mir210 which exclusively regulated by HIF.

The EPC response will be evaluated at the same time points by Fluorescence-activated Cell Sorting (FACS) analysis of the number of Hematopoietic progenitor cell antigen (CD34+)/ CD133 antigen/Kinase insert domain receptor (KDR +)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type1 diabetes with a duration of the disease between 10-20 years (HbA1c ≥ 55 mmol/mol)
2. Age 18-55
3. Diabetes duration 5-40 years
4. Contraception: Female subjects must be postmenopausal, surgically sterile, or if premenopausal (and not surgically sterile), be prepared to use more than 1 effective method of contraception during the study and for 30 days after the last visit. Effective methods of contraception are considered to be those listed below:

   1. Double barrier method, i.e. (a) condom (male or female) or (b) diaphragm, with spermicide; or
   2. Intrauterine device; or
   3. Vasectomy (partner); or
   4. Hormonal (e.g. contraceptive pill, patch, intramuscular implant or injection); or
   5. Abstinence, if in line with the preferred and usual lifestyle of the subject.
5. Signed informed consent

Exclusion Criteria:

1. Smoking
2. Infections during the last month
3. Major cardiovascular complications such as coronary heart disease, unstable or stable angina, myocardial infarction, ventricular arrhythmias, and atrial fibrillation in the last 3 months
4. Decompensated congestive heart failure or functional class 3-4.
5. therapy with beta-blockers
6. severe hypertension (180 mmHg systolic or 110 mmHg diastolic blood pressure
7. proliferative retinopathy.
8. Sign for peripheral diabetic neuropathy (decreased/absent sensitivity to 10 g monofilament, vibration, plantar reflex)
9. definite autonomic dysfunction
10. HbA1c > 100 mmol/l
11. Any concomitant disease or condition that may interfere with the possibility for the patient to comply with or complete the study protocol
12. Malignancy
13. History of alcohol or drug abuse
14. Participant in another ongoing pharmacological study
15. If female: plans to become pregnant, known pregnancy or a positive urine pregnancy test (confirmed by a positive serum pregnancy test), or lactating
16. Unwillingness to participate following oral and written information
17. Subjects with any other severe acute or chronic medical or psychiatric condition that make the subject inappropriate for the study in the judgment of the investigator
18. History of anemia, bleeding gastric ulcer, abundant menstruation
19. Treatment with prochlorperazine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-12-12 (Estimated); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
Endothelial precursor cell account (EPC) | 24 hours
  The absolute amount of endothelial precursor cells in 10 ml of blood

CONTACTS AND LOCATIONS:
Overall Officials: Sergiu Catrina, Ass. prof., Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arden GB, Sivaprasad S. The pathogenesis of early retinal changes of diabetic retinopathy. Doc Ophthalmol. 2012 Feb;124(1):15-26. doi: 10.1007/s10633-011-9305-y. PMID 22302291
- [Background] Schaper NC, Huijberts M, Pickwell K. Neurovascular control and neurogenic inflammation in diabetes. Diabetes Metab Res Rev. 2008 May-Jun;24 Suppl 1:S40-4. doi: 10.1002/dmrr.862. PMID 18442183
- [Background] Flyvbjerg A. Diabetic angiopathy, the complement system and the tumor necrosis factor superfamily. Nat Rev Endocrinol. 2010 Feb;6(2):94-101. doi: 10.1038/nrendo.2009.266. PMID 20098449
- [Background] Ruiter MS, van Golde JM, Schaper NC, Stehouwer CD, Huijberts MS. Diabetes impairs arteriogenesis in the peripheral circulation: review of molecular mechanisms. Clin Sci (Lond). 2010 Jun 8;119(6):225-38. doi: 10.1042/CS20100082. PMID 20545627
- [Background] Friederich M, Fasching A, Hansell P, Nordquist L, Palm F. Diabetes-induced up-regulation of uncoupling protein-2 results in increased mitochondrial uncoupling in kidney proximal tubular cells. Biochim Biophys Acta. 2008 Jul-Aug;1777(7-8):935-40. doi: 10.1016/j.bbabio.2008.03.030. Epub 2008 Apr 7. PMID 18439413
- [Background] Ivan M, Kondo K, Yang H, Kim W, Valiando J, Ohh M, Salic A, Asara JM, Lane WS, Kaelin WG Jr. HIFalpha targeted for VHL-mediated destruction by proline hydroxylation: implications for O2 sensing. Science. 2001 Apr 20;292(5516):464-8. doi: 10.1126/science.1059817. Epub 2001 Apr 5. PMID 11292862
- [Background] Elson DA, Ryan HE, Snow JW, Johnson R, Arbeit JM. Coordinate up-regulation of hypoxia inducible factor (HIF)-1alpha and HIF-1 target genes during multi-stage epidermal carcinogenesis and wound healing. Cancer Res. 2000 Nov 1;60(21):6189-95. PMID 11085544
- [Background] Ceradini DJ, Kulkarni AR, Callaghan MJ, Tepper OM, Bastidas N, Kleinman ME, Capla JM, Galiano RD, Levine JP, Gurtner GC. Progenitor cell trafficking is regulated by hypoxic gradients through HIF-1 induction of SDF-1. Nat Med. 2004 Aug;10(8):858-64. doi: 10.1038/nm1075. Epub 2004 Jul 4. PMID 15235597
- [Background] Devlin C, Greco S, Martelli F, Ivan M. miR-210: More than a silent player in hypoxia. IUBMB Life. 2011 Feb;63(2):94-100. doi: 10.1002/iub.427. Epub 2011 Feb 24. PMID 21360638
- [Background] Epstein AC, Gleadle JM, McNeill LA, Hewitson KS, O'Rourke J, Mole DR, Mukherji M, Metzen E, Wilson MI, Dhanda A, Tian YM, Masson N, Hamilton DL, Jaakkola P, Barstead R, Hodgkin J, Maxwell PH, Pugh CW, Schofield CJ, Ratcliffe PJ. C. elegans EGL-9 and mammalian homologs define a family of dioxygenases that regulate HIF by prolyl hydroxylation. Cell. 2001 Oct 5;107(1):43-54. doi: 10.1016/s0092-8674(01)00507-4. PMID 11595184
- [Background] Mehrabani M, Najafi M, Kamarul T, Mansouri K, Iranpour M, Nematollahi MH, Ghazi-Khansari M, Sharifi AM. Deferoxamine preconditioning to restore impaired HIF-1alpha-mediated angiogenic mechanisms in adipose-derived stem cells from STZ-induced type 1 diabetic rats. Cell Prolif. 2015 Oct;48(5):532-49. doi: 10.1111/cpr.12209. PMID 26332145
- [Background] Weng R, Li Q, Li H, Yang M, Sheng L. Mimic hypoxia improves angiogenesis in ischaemic random flaps. J Plast Reconstr Aesthet Surg. 2010 Dec;63(12):2152-9. doi: 10.1016/j.bjps.2010.02.001. Epub 2010 Mar 31. PMID 20359971
- [Background] Botusan IR, Sunkari VG, Savu O, Catrina AI, Grunler J, Lindberg S, Pereira T, Yla-Herttuala S, Poellinger L, Brismar K, Catrina SB. Stabilization of HIF-1alpha is critical to improve wound healing in diabetic mice. Proc Natl Acad Sci U S A. 2008 Dec 9;105(49):19426-31. doi: 10.1073/pnas.0805230105. Epub 2008 Dec 4. PMID 19057015
- [Background] Catrina SB. Impaired hypoxia-inducible factor (HIF) regulation by hyperglycemia. J Mol Med (Berl). 2014 Oct;92(10):1025-34. doi: 10.1007/s00109-014-1166-x. Epub 2014 Jun 12. PMID 25027070
- [Background] Ram M, Singh V, Kumawat S, Kumar D, Lingaraju MC, Uttam Singh T, Rahal A, Kumar Tandan S, Kumar D. Deferoxamine modulates cytokines and growth factors to accelerate cutaneous wound healing in diabetic rats. Eur J Pharmacol. 2015 Oct 5;764:9-21. doi: 10.1016/j.ejphar.2015.06.029. Epub 2015 Jun 19. PMID 26101070
- [Background] Wang C, Cai Y, Zhang Y, Xiong Z, Li G, Cui L. Local injection of deferoxamine improves neovascularization in ischemic diabetic random flap by increasing HIF-1alpha and VEGF expression. PLoS One. 2014 Jun 25;9(6):e100818. doi: 10.1371/journal.pone.0100818. eCollection 2014. PMID 24963878
- [Background] Hou Z, Nie C, Si Z, Ma Y. Deferoxamine enhances neovascularization and accelerates wound healing in diabetic rats via the accumulation of hypoxia-inducible factor-1alpha. Diabetes Res Clin Pract. 2013 Jul;101(1):62-71. doi: 10.1016/j.diabres.2013.04.012. Epub 2013 May 28. PMID 23726275
- [Background] Smith TG, Balanos GM, Croft QP, Talbot NP, Dorrington KL, Ratcliffe PJ, Robbins PA. The increase in pulmonary arterial pressure caused by hypoxia depends on iron status. J Physiol. 2008 Dec 15;586(24):5999-6005. doi: 10.1113/jphysiol.2008.160960. Epub 2008 Oct 27. PMID 18955380
- [Background] Ren X, Dorrington KL, Maxwell PH, Robbins PA. Effects of desferrioxamine on serum erythropoietin and ventilatory sensitivity to hypoxia in humans. J Appl Physiol (1985). 2000 Aug;89(2):680-6. doi: 10.1152/jappl.2000.89.2.680. PMID 10926654
- [Background] Balanos GM, Dorrington KL, Robbins PA. Desferrioxamine elevates pulmonary vascular resistance in humans: potential for involvement of HIF-1. J Appl Physiol (1985). 2002 Jun;92(6):2501-7. doi: 10.1152/japplphysiol.00965.2001. PMID 12015365
- [Background] Duennwald T, Bernardi L, Gordin D, Sandelin A, Syreeni A, Fogarty C, Kyto JP, Gatterer H, Lehto M, Horkko S, Forsblom C, Burtscher M, Groop PH; FinnDiane Study Group. Effects of a single bout of interval hypoxia on cardiorespiratory control in patients with type 1 diabetes. Diabetes. 2013 Dec;62(12):4220-7. doi: 10.2337/db13-0167. Epub 2013 Jun 3. PMID 23733200
- [Background] Duennwald T, Gatterer H, Groop PH, Burtscher M, Bernardi L. Effects of a single bout of interval hypoxia on cardiorespiratory control and blood glucose in patients with type 2 diabetes. Diabetes Care. 2013 Aug;36(8):2183-9. doi: 10.2337/dc12-2113. Epub 2013 Mar 27. PMID 23536585
- [Background] Balczewska D, Ptaszynski P, Cygankiewicz I. [Baroreflex sensitivity: measurement and clinical aspects]. Przegl Lek. 2015;72(11):682-9. Polish. PMID 27012131
- [Background] Svacinova J, Moudr J, Honzikova N. [Baroreflex sensitivity: diagnostic importance, methods of determination and a model of baroreflex blood-pressure regulation]. Cesk Fysiol. 2013;62(1):10-8. Czech. PMID 23821958
- [Background] Collier DJ, Bernardi L, Angell-James JE, Caulfield MJ, Sleight P; Anglo-Scandinavian Cardiac Outcomes Trial. Baroreflex sensitivity and heart rate variability as predictors of cardiovascular outcome in hypertensive patients with multiple risk factors for coronary disease. J Hum Hypertens. 2001 Aug;15 Suppl 1:S57-60. doi: 10.1038/sj.jhh.1001077. No abstract available. PMID 11685912
- [Background] La Rovere MT, Maestri R, Robbi E, Caporotondi A, Guazzotti G, Febo O, Pinna GD. Comparison of the prognostic values of invasive and noninvasive assessments of baroreflex sensitivity in heart failure. J Hypertens. 2011 Aug;29(8):1546-52. doi: 10.1097/HJH.0b013e3283487827. PMID 21666492